CLINICAL TRIAL: NCT05551520
Title: ImPACT Version 4-Touchscreen: Normative and Reliability Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ImPACT Applications, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: QPR-21-20
Record Dates: First submitted 2022-03-29; First posted 2022-09-22 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Concussion
Keywords: Brain
MeSH Terms: conditions — Brain Concussion | interventions — Reproducibility of Results

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Normative (Other): ImPACT will be administered to participant's for a baseline test.
  Interventions: Device: Normative
- Reliability (Other): ImPACT will be administered to participant's within 60 days of baseline test.
  Interventions: Device: Reliability

INTERVENTIONS:
Device: Normative — ImPACT will be administered at baseline testing
  Arms: Normative
Device: Reliability — ImPACT will be administered again within 60 days of baseline test
  Arms: Reliability

SUMMARY:
This research study is designed to establish normative database and reliability of ImPACT for adolescents and adults ages 12 through 80 to expand the use of devices to include touchscreen.

DETAILED DESCRIPTION:
This research study is designed to establish normative database and reliability of ImPACT for adolescents and adults ages 12 through 80 to expand the use of devices to include touchscreen. Enrollment will be 900 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-80
2. Primary English speaking or fluent in English

Exclusion Criteria:

1. Documentation of a known special education diagnosis other than a 504 designation.
2. History of concussion less than 6 months to the study participation
3. Known physical (e.g., visual impairment not fixable by usual means, such as glasses) or psychological impairment (ADHD, LDD, etc.) that would affect their ability to perform the test.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1437 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Validity | 12 months
  ImPACT Touchscreen performs within normal parameters of ImPACT Online

SECONDARY OUTCOMES:
Reliability | Baseline test will be administered at enrollment and re-test will be administered within 60 days of baseline test.
  Reliability will be established through a test/re-test. ImPACT Touchscreen will be administered at 2 time points to establish results should be stable over time.

CONTACTS AND LOCATIONS:
Locations (1):
- ImPACT Applications, Inc., Coralville, Iowa, United States